CLINICAL TRIAL: NCT06260098
Title: StressLess Yoga Study: A Scientific Exploration of Yoga for Stress Reduction
Brief Title: StressLess Yoga Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Crystal Park, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H23-0617
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stress
MeSH Terms: interventions — Yoga; Meditation; Posture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga with High Breath work & meditation; Low movement/postures (Experimental)
  Interventions: Behavioral: Yoga with High Breath work & meditation; Low movement/postures
- Yoga with Low Breath work & meditation; High movement/postures (Experimental)
  Interventions: Behavioral: Yoga with Low Breath work & meditation; High movement/postures

INTERVENTIONS:
Behavioral: Yoga with High Breath work & meditation; Low movement/postures — Participants will engage in an 8 week asynchronous yoga class focused on the internal and cognitive experience within the practice using breathing and meditation focused techniques.
  Arms: Yoga with High Breath work & meditation; Low movement/postures
Behavioral: Yoga with Low Breath work & meditation; High movement/postures — Participants will engage in an 8 week asynchronous yoga class with a emphasis on the physicality and movements of the practice.
  Arms: Yoga with Low Breath work & meditation; High movement/postures

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of using an asynchronous online yoga program to reduce stress. The study will use an 8 week asynchronous yoga intervention of two different types of yoga (high in breath work and meditation; low in vigorous movement/postures vs. low breath work and meditation; high movement/postures). In addition to self-report stress, measures include sleep, heart rate variability, mindfulness, Essential Properties of Yoga, and acceptability questions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Self-identification as "stressed"
* Scoring 8 or higher on the Perceived Stress Scale (PSS) indicating moderate-to-high stress
* Willingness to complete the 8-week yoga intervention
* Willingness to attend baseline and follow-up visits
* Ability to read and write in English
* Having practiced yoga ≤ 2x in the last 6 months

Exclusion Criteria:

* Serious or unstable psychiatric illness (e.g., psychosis, mania)
* Major coexisting medical illness (e.g., cancer, COPD, obesity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
The number (percentage)of people completing the whole protocol (6/8 yoga classes & 2 in-person visits) | 8 weeks
  The number (percentage)of people completing the whole protocol (6/8 yoga classes & 2 in-person visits)
The combined score (out of 35) on the 5-item Treatment Acceptability Questionnaire (TAQ) | 8 weeks
  The combined score (out of 35) on the 5-item Treatment Acceptability Questionnaire (TAQ). The measure is scored on a 1-7 Likert scale. Higher scores indicate highly acceptable, ethical, knowledgeable, and trustworthy study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Bousfield Psychology Building, 406 Babbidge Road, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No